CLINICAL TRIAL: NCT07226440
Title: Assessing the Impact of a Bile Acid Sequestrant on Serum PFAS Levels in Highly Exposed Individuals
Brief Title: Examining a Novel Gastrointestinal Intervention to Negate Environmental Toxicants (ENGINE)
Acronym: ENGINE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ENGINE-01
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Toxicant Exposure; Firefighter; Occupational Exposure to Chemicals
Keywords: Per- and polyfluoroalkyl substances; PFAS; Firefighters; Occupational exposure; Bile acid sequestrants; Colesevelam
MeSH Terms: conditions — Progressive Encephalomyelitis with Rigidity | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, crossover trial with a 2-week washout between treatment periods. Participants are assigned to one of two sequences: colesevelam followed by placebo, or placebo followed by colesevelam.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All study staff will be masked. The only unmasked individuals will be the pharmacists dispensing in the medication/placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colesevelam first (Active Comparator): Participants randomized to this arm will receive colesevelam, taking 3 tablets twice daily for 12 weeks, followed by a 2-week washout period, and then 12 weeks of matching placebo tablets taken on the same schedule. Both the study drug and the placebo will be provided in identical-appearing bottles to maintain blinding.
  Interventions: Drug: Colesevelam; Drug: Placebo
- Placebo first (Placebo Comparator): Participants randomized to this arm will receive placebo tablets, taking 3 tablets twice daily for 12 weeks, followed by a 2-week washout period, and then 12 weeks of colesevelam (3 tablets twice daily). Both the study drug and the placebo will be provided in identical-appearing bottles to maintain blinding.
  Interventions: Drug: Colesevelam; Drug: Placebo

INTERVENTIONS:
Drug: Colesevelam — Colesevelam in 625-mg tablets. Participants will take 3 tablets orally, twice daily (total daily dose 3.75 g) for 12 weeks.
  Other Names: Welchol
Drug: Placebo — Matching inert oral tablets designed to mimic colesevelam 625 mg tablets in size, shape, and color, but containing no active pharmaceutical ingredient. Participants will take 3 orally, twice per day for 12 weeks.
  Other Names: Inert oral tablets

SUMMARY:
This randomized, placebo-controlled crossover trial will test the feasibility and acceptability of using colesevelam in male firefighters with high per- and polyfluoroalkyl substances (PFAS) exposure. This trial will also explore whether colesevelam lowers blood PFAS levels and urine environmental toxicant and mold mycotoxin levels.

DETAILED DESCRIPTION:
Firefighters experience elevated exposure to per- and polyfluoroalkyl substances (PFAS) through firefighting foams, turnout gear, and dust in fire stations. PFAS persist in the body due to their long biological half-lives, leading to bioaccumulation and raising concern for adverse effects on hormone regulation, immune function, reproduction, and cancer risk. Despite growing awareness, there are no approved treatment options to reduce PFAS levels in humans. Bile acid sequestrants, such as colesevelam, bind bile acids in the gastrointestinal tract and may interrupt enterohepatic recirculation of PFAS, thereby enhancing elimination. Observational studies and one small randomized trial suggest that bile acid sequestrants can meaningfully reduce PFAS levels. This trial will evaluate the feasibility, adherence, and acceptability of colesevelam in male firefighters with elevated PFAS, while exploring its effects on serum PFAS concentrations and urine environmental toxicant and mold mycotoxin levels.

ELIGIBILITY:
Inclusion Criteria:

* Male firefighter
* California resident
* Age 18-64
* Full-time, active-duty (fire suppression and/or arson investigation)
* English-speaking
* Access to a reliable internet connection
* Willing to attend 3 in-person study visits in the San Francisco Bay Area over about 6.5 months
* Willing to receive weekly text message reminders to complete online surveys
* Willing to complete a mail-based, at-home finger-prick blood test
* Willing to take 3 tablets (each tablet about the size of a multivitamin) orally twice daily for a total of 6 months
* Evaluated by study team to have an elevated risk of PFAS exposure (e.g., duration of firefighting service, prior NASEM-7 result greater than or equal to 10)

Exclusion Criteria:

* Gastroparesis or other severe gastrointestinal motility disorders
* Bowel obstruction
* History of major gastrointestinal tract surgery
* Dysphagia or difficulty swallowing (due to tablet size)
* History of hypertriglyceridemia (triglycerides exceeding 500 mg/dL)
* History of hypertriglyceridemia-induced pancreatitis
* Type 1 or 2 diabetes
* History of fat-soluble vitamin deficiencies i.e., vitamins A, D, E, or K
* Phenylketonuria
* History of known bleeding/clotting disorders
* Medications or treatments that may impact the excretion of PFAS, such as activated charcoal, other bile acid sequestrants, chelation therapies, etc.
* More than one blood or plasma donation in the past 12 months and/or unalterable plans to donate blood or plasma during the study participation period
* Use of clomiphene, testosterone, human chorionic gonadotropin, anabolic steroids, anastrozole or any other substances that may impact testosterone levels in males

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Retention | Enrollment to Week 27
  Proportion completing all study blood draws after consent
Adherence to study drug | Enrollment to Week 27
  Proportion taking ≥80% of colesevelam doses
Adherence to placebo | Enrollment to Week 27
  Proportion taking ≥80% of placebo doses
Acceptability | Week 27
  Proportion endorsing "likely" or "very likely" to refer a co-worker to the study
Likability | Week 27
  Proportion endorsing "likely" or "very likely" to participate again

SECONDARY OUTCOMES:
Serum PFAS Levels | Baseline (Week 0) to the end of each 12-week intervention period (Weeks 13 and 27)
  Between-period and within-person changes in serum concentrations of the National Academy of Sciences, Engineering, and Medicine (NASEM)-7 PFAS score (sum of seven PFAS analytes). Higher scores mean higher PFAS levels in the body. Scores range from 0 to an unknown maximum.

OTHER OUTCOMES:
Urine Mold Mycotoxin Levels | Baseline (Week 0) to the end of each 12-week intervention period (Weeks 13 and 27)
  Between-period and within-person changes in urine concentrations of mold mycotoxins
Urine Environmental Toxicant Levels | Baseline (Week 0) to the end of each 12-week intervention period (Weeks 13 and 27)
  Between-period and within-person changes in urine concentrations of environmental toxicants

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California San Francisco, Osher Center for Integrative Health; Leena Pandya, ND, Principal Investigator — University of California San Francisco, Osher Center for Integrative Health; Sarah Fisher, MS, Study Director — University of California San Francisco, Osher Center for Integrative Health
Locations (1):
- UCSF Osher Center for Integrative Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigative team will share de-identified data, an associated codebook, and an abbreviated study protocol.
Supporting Information: Study Protocol, ICF
Time Frame: The investigative team will share data one year after all study participants' participation has concluded.
Access Criteria: The investigative team will make data accessible via an online data sharing repository
URL: https://osf.io

REFERENCES:
- [Background] Johnson JD, Gibson SJ, Ober RE. Cholestyramine-enhanced fecal elimination of carbon-14 in rats after administration of ammonium [14C]perfluorooctanoate or potassium [14C]perfluorooctanesulfonate. Fundam Appl Toxicol. 1984 Dec;4(6):972-6. doi: 10.1016/0272-0590(84)90235-5. PMID 6519377
- [Background] Mazumder NU, Hossain MT, Jahura FT, Girase A, Hall AS, Lu J, Ormond RB. Firefighters' exposure to per-and polyfluoroalkyl substances (PFAS) as an occupational hazard: A review. Front Mater. 2023;10:10.3389/fmats.2023.1143411. doi: 10.3389/fmats.2023.1143411. Epub 2023 Mar 23. PMID 38074949
- [Background] Young AS, Sparer-Fine EH, Pickard HM, Sunderland EM, Peaslee GF, Allen JG. Per- and polyfluoroalkyl substances (PFAS) and total fluorine in fire station dust. J Expo Sci Environ Epidemiol. 2021 Sep;31(5):930-942. doi: 10.1038/s41370-021-00288-7. Epub 2021 Feb 5. PMID 33542478
- [Background] Lucas K, Gaines LGT, Paris-Davila T, Nylander-French LA. Occupational exposure and serum levels of per- and polyfluoroalkyl substances (PFAS): A review. Am J Ind Med. 2023 May;66(5):379-392. doi: 10.1002/ajim.23454. Epub 2022 Dec 27. PMID 36573587
- [Background] Moller JJ, Lyngberg AC, Hammer PEC, Flachs EM, Mortensen OS, Jensen TK, Jurgens G, Andersson A, Soja AMB, Lindhardt M. Substantial decrease of PFAS with anion exchange resin treatment - A clinical cross-over trial. Environ Int. 2024 Mar;185:108497. doi: 10.1016/j.envint.2024.108497. Epub 2024 Feb 13. PMID 38367552
- [Background] Ducatman A, Luster M, Fletcher T. Perfluoroalkyl substance excretion: Effects of organic anion-inhibiting and resin-binding drugs in a community setting. Environ Toxicol Pharmacol. 2021 Jul;85:103650. doi: 10.1016/j.etap.2021.103650. Epub 2021 Apr 2. PMID 33819618
- [Background] Seyyedsalehi MS, Boffetta P. Per- and Poly-fluoroalkyl Substances (PFAS) Exposure and Risk of Kidney, Liver, and Testicular Cancers: A Systematic Review and Meta-Analysis. Med Lav. 2023 Oct 24;114(5):e2023040. doi: 10.23749/mdl.v114i5.15065. PMID 37878255